CLINICAL TRIAL: NCT07133009
Title: The Effect of the Intentional Relationship Model on Therapeutic Use of Self and Career Choice in Occupational Therapy Students
Brief Title: Intentional Relationship Model in OT Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Medipol University (Other)
Responsible Party: Principal Investigator, Busra Kaplan Kilic, Assist Prof, Ankara Medipol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: E-2025-08-01; Busra Kaplan Kilic (Other: Ankara Medipol University)
Record Dates: First submitted 2025-08-01; First posted 2025-08-20 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-10

CONDITIONS: Occupational Therapy Students
Keywords: Vocational Choice; Therapeutic Use of Self; Intentional Relationship Model; Occupational Therapy Students

STUDY DESIGN:
Intervention Model Description: There is no control group in this study. Data collection tools will be applied before and after training in a single group.
Masking Description: Participants and researchers have been informed about the study. However, assistance will be sought from an independent evaluator who has not been informed about the study regarding the analysis of the outcome measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training Group (Other): Participants will undergo an IRM-based training program. Based on the IRM model, the six-week training program will consist of 30 minutes of theoretical instruction on a designated topic each week, followed by 30 minutes of role-playing scenarios related to the topic covered.
  Interventions: Other: Intentional Relationship Model (IRM) Training

INTERVENTIONS:
Other: Intentional Relationship Model (IRM) Training — 1 Theory: Brief introduction to the Intentional Relationship Model, therapeutic self-awareness, and explanation of therapeutic styles.
  1. Practice: Students share their existing knowledge and thoughts about therapeutic styles, and discuss the practical implications of therapeutic styles that may be relevant to them.
  2. Theory: Information about defining interpersonal characteristics and getting to know our clients
  2 Practice: Sources of differences in client profiles in the client-therapist relationship, structuring questions appropriately, and practices for getting to know our clients better 3 Theory: Information about potential difficulties that may arise in the therapeutic process 3 Practice: Scenarios are played out about what can be done to address difficulties that may arise in the client-therapist relationship 4 Theory: Information about interpersonal reasoning skills and coping with difficulties 4 Practice: Strategies that can be used to create an appropriat

SUMMARY:
This study aims to examine the changes in occupational therapy interns' professional personality types and therapeutic use behaviors through an Intentional Relationship Model (IRM)-based training program. The study aims to introduce a therapeutic relationship-focused approach to occupational therapy education and to contribute to the effective development of students' therapeutic use skills during their professional development process.

Participants will receive one hour of interactive training per week for six weeks, structured within the framework of the IRM.

DETAILED DESCRIPTION:
Type of research: Cross-sectional research Population and sample: The population of the research will consist of volunteer occupational therapy 4th grade students. In order to determine the sample size, a power analysis was conducted using the G*Power program with 95% power (alpha=0.05, two-tailed), and it was determined that a minimum of 54 participants were required for a matched t-test based on the guidelines provided by Cohen.

Inclusion criteria:

* Being a 4th-year occupational therapy student
* Being literate in Turkish

Exclusion criteria:

● Not participating regularly in the education program Students who meet the participation criteria and are provided with detailed information about the study will be asked to sign an informed consent form if they voluntarily agree to participate in the study. While the assessments will be conducted face-to-face, the education program will be conducted online (via Zoom).

Forms used for data collection: Sociodemographic Form, Self-Efficacy for Therapeutic Use of Self (SETUS), Holland's Vocational Choice There is no control group in this study. Data collection tools will be applied before and after training in a single group.

ELIGIBILITY:
Inclusion Criteria:

* Be a 4th-year student in the Occupational Therapy Department,
* Be an intern student,
* Be literate in Turkish

Exclusion Criteria:

* Failure to attend the training program regularly
* Having a chronic illness

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Self-Efficacy for Therapeutic Use of Self Scale (SETUS) | It will be administered to each participant before the training and six weeks after the training is completed.
  This tool based on a combination of Bandura's social cognitive theory and Taylor's model of the therapeutic relationship in occupational therapy (IRM). The SETUS instrument measures therapists' self-efficacy in three different aspects of therapeutic use of self, according to Taylor's outline in the IRM of the essential aspects of relating in therapeutic contexts. The first 6 items of the SETMU, 7-18th of the SERIC, and 19-20th of the SEMIE subscale items form the whole scale SETUS. The items in the scale were related to occupational therapists' competencies in using therapeutic use of self while working with their clients. Ten Likert-type scales were used, such as I cannot do it at all (1point), I can do it moderately (6 point), and I can definitely do it (10 point). A high score indicates high self-efficacy in therapeutic use of self.

SECONDARY OUTCOMES:
Holland Vocational Preference Inventory | It will be administered to each participant before the training and six weeks after the training is completed.
  Holland proposed that people can be divided into six groups based on their personality traits and that these six groups can be grouped in the same way in their professional environments. Based on this, he developed the Personality Theory, known as the Typology Theory, in the field of career counseling. The main objective of this theory is to explain individuals' professional behaviors and to make recommendations for them to achieve professional satisfaction when choosing or changing careers. For the analysis of personality types, Holland's Career Preference Inventory included 90 questions to identify each personality type. The responses were coded using a 3-point Likert scale: "2 = I like it," "1 = It doesn't matter," and "0 = I don't like it." Scoring was based on participants' responses to determine the personality types they were closest to and farthest from.

CONTACTS AND LOCATIONS:
Overall Officials: Busra Kaplan Kilic, PhD, Principal Investigator — Ankara Medipol University
Locations (1):
- Ankara Medipol University, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yazdani F, Carstensen T, Bonsaksen T. Therapeutic mode preferences and associated factors among Norwegian undergraduate occupational therapy students: A cross-sectional exploratory study. Scand J Occup Ther. 2017 Mar;24(2):136-142. doi: 10.1080/11038128.2016.1220620. Epub 2016 Aug 19. PMID 27538471
- [Background] Schwank K, Carstensen T, Yazdani F, Bonsaksen T. The Course of Self-Efficacy for Therapeutic Use of Self in Norwegian Occupational Therapy Students: A 10-Month Follow-Up Study. Occup Ther Int. 2018 Apr 1;2018:2962747. doi: 10.1155/2018/2962747. eCollection 2018. PMID 29805333